CLINICAL TRIAL: NCT03508843
Title: Improving Child Restraint Installation in Rural America Through Interactive Virtual Presence
Brief Title: Improving Child Restraint Installation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Schwebel, University Professor & Associate Dean, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 300001220
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Car Seat Installation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interactive virtual presence (Experimental): install a car seat using advice from a remotely-located certified car seat technician communicating via interactive virtual presence
  Interventions: Behavioral: interactive virtual presence

INTERVENTIONS:
Behavioral: interactive virtual presence — installing the car seat with advice via interactive virtual presence

SUMMARY:
The investigators will conduct a pre-post trial with 150 parents in rural South Central Montana. The study will recruit families to cooperating community locations (e.g., churches, public libraries) to participate in research evaluating the efficacy of parents installing restraints with guidance from a remotely-located technician using interactive virtual presence. Following informed consent procedures, parents will complete a brief survey on behaviors, attitudes, and perceptions about child safety and restraints while an on-site technician evaluates baseline safety of the restraint. Parents will then engage remotely using their personal smartphone with an off-site certified car seat technician, obtaining advice to install the child restraint properly via the HelpLightning interactive virtual presence app. Following the remote interaction, the on-site technician will again inspect the restraint using the validated checklist (and correct any errors prior to the participant leaving). The overall goal is to demonstrate installation of child restraints can be effectively accomplished to rural populations using interactive virtual presence. The study has 2 specific aims:

Specific Aim 1. Demonstrate technological and behavioral efficacy of providing instructions on child restraint installation remotely to rural populations. Demonstrate >95% of interactions proceed without technical problems, without reports of communication difficulty on either end of the exchange (the parent or the technician), and without interruption.

Specific Aim 2. Identify accuracy of child restraint installation by parents using instructions provided by a remotely-located certified technician via interactive virtual presence. Demonstrate installation in this manner achieves ≥90% accuracy across all aspects of child restraint installation. Demonstrate installation in this manner significantly reduces restraint installation errors.

ELIGIBILITY:
Inclusion Criteria:

* communicate in English
* drive a vehicle with one or more car seats present
* willing to install a car seat into the vehicle

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Schwebel, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interactive Virtual Presence
Started | 150
Completed | 147
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — technical difficulties | 2

BASELINE CHARACTERISTICS:
Population: Adult caregivers of young children from southeast Montana who drove a vehicle with a child restraint in it. Participants for whom <70% of items in a category could be coded at baseline or post-intervention were excluded from those analyses; common exclusions were baseline situations with uninstalled restraint or children not present.
Arm/Group | Interactive Virtual Presence
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 137
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 111
  More than one race | 0
  Unknown or Not Reported | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Accurately Select a Safe Child Restraint
Description: accurate selection of a safe child restraint that was proper for the child's age and size
Time Frame: immediately (< 5 minutes) after the car seat is installed
Population: comparison to baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Virtual Presence
Number analyzed (Participants) | 142
Participants
  post-intervention | 131
  baseline | 121
Statistical Analysis 1: Comparison: Interactive Virtual Presence; Test type: Superiority; p < .001, McNemar

2. Primary Outcome: Number of Participants Who Install the Child Restraint Accurately Into the Vehicle
Description: accurate installation of the child restraint into the vehicle
Time Frame: immediately (< 5 minutes) after the car seat is installed
Population: comparison to baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Virtual Presence
Number analyzed (Participants) | 120
Participants
  post-intervention | 45
  baseline | 18
Statistical Analysis 1: Comparison: Interactive Virtual Presence; Test type: Superiority; p < .001, McNemar

3. Primary Outcome: Number of Participants Who Properly Position the Child Restraint in the Vehicle
Description: proper positioning of the child restraint in the vehicle
Time Frame: immediately (< 5 minutes) after the car seat is installed
Population: comparison to baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Virtual Presence
Number analyzed (Participants) | 77
Participants
  post-intervention | 51
  baseline | 33
Statistical Analysis 1: Comparison: Interactive Virtual Presence; Test type: Superiority; p > .05, McNemar

ADVERSE EVENTS:
Time Frame: 45 minutes, from baseline through post-intervention assessment
Arm/Group | Interactive Virtual Presence
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03508843/Prot_SAP_000.pdf